CLINICAL TRIAL: NCT01930747
Title: Impact of Deep Neuromuscular Block Versus Inhalation and Total Intravenous Anesthesia (TIVA) on Laparoscopic Surgical Workspace Defined as Insufflated Pneumoperitoneum Volume.
Brief Title: Effect of Deep Neuromuscular Block (NMB), Inhalation or TIVA on Pneumoperitoneum.
Acronym: TIVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Jan Paul J Mulier MD PhD, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013JPM2
Record Dates: First submitted 2013-05-30; First posted 2013-08-29 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Muscle Relaxation
Keywords: pneumoperitoneum; laparoscopy
MeSH Terms: conditions — Pneumoperitoneum | interventions — Rocuronium; Sevoflurane; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- deep neuromuscular block (Experimental): deep neuromuscular block is given after first measurement of lap workspace one bolus dose of 1 mg/kg rocuronium is given
  Interventions: Drug: rocuronium
- inhalation with 1 MAC Sevoflurane (Experimental): 1 MAC Sevoflurane inhalation is given after first measurement of lap workspace
  Interventions: Drug: Sevoflurane
- remifentanyl (Experimental): remifentanyl infusion is given after first measurement of lap workspace
  Interventions: Drug: remifentanyl

INTERVENTIONS:
Drug: rocuronium — measure effect on laparoscopic workspace
  Other Names: esmeron
  Arms: deep neuromuscular block
Drug: Sevoflurane — 1 MAC sevoflurane inhalation is given
  Other Names: sevorane
  Arms: inhalation with 1 MAC Sevoflurane
Drug: remifentanyl — remifentanyl is given in infusion
  Other Names: ultiva
  Arms: remifentanyl

SUMMARY:
The objective of this study is to compare the value of deep neuromuscular block (NMB) (using rocuronium) in laparoscopy versus high dose opioids (using remifentanil) or 1 minimum alveolar concentration (MAC) inhalation (using sevoflurane) for the surgeon.

The study hypothesis is that laparoscopic workspace is larger when using rocuronium versus opioids or inhalation. Laparoscopic workspace is measured as the abdominal compliance and the pressure at volume zero (PV0) using the abdominal pressure volume relation. Three points allow to calculate the abdominal compliance and the pressure at zero volume (PV0).

DETAILED DESCRIPTION:
Background and rationale

The value of administering a deep neuromuscular block (NMB) to reach a post-tetanic count (PTC) of < 4 during laparoscopy is not clear. Some anesthesiologists claim that certain laparoscopic procedures do not need NMB at all and that surgeons cannot objectivize the existence of insufficient workspace and the effect of NMB. They assume that deep anesthesia with remifentanyl improves also the workspace. This assumption may be based on the fact that deep anesthesia prevents spontaneous active muscle contractions. However, preventing an active contraction through deep anesthesia is different from blocking the "active tonus" with a NMB.

Due to the difficulties in evaluating the surgical access, surgical workspace (1) should be measured as the inflated carbon dioxide (CO2) volume for a given intra-abdominal pressure during pneumoperitoneum. Abdominal compliance (C or its reciprocal the elastance: E) and the pressure at zero volume (PV0) are calculated by measuring three or more pressure volume points to construct the abdominal pressure volume relation.

The objective of this study is to compare the value of deep NMB (using rocuronium) in laparoscopy versus high dose opioids (using remifentanil) or 1 Minimum alveolar concentration (MAC) inhalation (using sevoflurane) for the surgeon.

Objectives

1. Primary Efficacy Objective: To compare the impact of the following agents on the reduction in active muscle tonus during laparoscopy (time frame: during surgery beig maximum 90 minutes) : remifentanyl > 0.50 µg/kg/min; sevoflurane > 1 MAC and deep neuromuscular block (rocuronium given with PTC < 4).
2. Primary Safety Objective: To compare the adverse events ( time frame: during hospitalisation maximum 3 days after surgery) among the patient groups who receive the different agents listed above in the "primary efficacy objective,"

Hypothesis

1. High dose remifentanyl does not increase laparoscopic surgical workspace compared to deep NMB (PTC < 4).
2. 1 MAC inhalation with sevoflurane does not increase laparoscopic surgical workspace compared to deep NMB ( PTC < 4)
3. Surgeons will encounter more workspace problems when no NMB is used.

Study design

Open randomized blinded clinical trial including:

1. Laparoscopic bariatric surgery in a patient older than 18 years of age without previous laparotomy. Examples of laparoscopic bariatric procedures are gastric band, sleeve gastrectomy, gastric bypass, gastric bypass after lap band, and revision of a gastric bypass.

and excluding:

1. Allergies or contraindications to the use of one or more of the following drugs: propofol, rocuronium, sugammadex, remifentanyl, or sevoflurane.
2. History of a laparotomy.
3. Emergency laparoscopy.

Methods:

Written informed consent will be obtained. The following patient characteristics will be noted: body weight, length, body mass index, age, sex, previous laparoscopic surgery, and gravidity for woman.

Anesthesia will be induced in all patients with Propofol 3 mg/kg ideal body weight (IBW), Ketamine 0,25 mg/kg IBW, Dexmedetomidine 1 ug/kg IBW loading dose, Lidocaine 1,5 mg/kg IBW and Succinylcholine 1 mg/kg total body weight (TBW).

Three Syringes with drugs (I II III) used in all patients (no investigation drugs):

I: Ketamine 50 mg (1cc); Lidocaine 300 mg (2% 15 cc), Dexmedetomidine 200 ug (1cc), 3 cc NaCl 0,9% in 20 cc syringe.

II: Propofol (10 mg/ml) not diluted in 50 cc syringe. III: Succinylcholine 200 mg (4cc) 16 cc NatriumChloride (NaCl) 0,9% in 20 cc syringe. (10 mg/ml)

Induction:

I: 1 ml/10 kg IBW II: 3 mg/ kg IBW or 3 ml/10 kg IBW III: 1 mg/kg TBW or 1ml /10 kg TBW

Maintenance:

I: 1 ml/10 kg IBW/ h. II: 0,5 tot 1 ml/ kg IBW/ h

Syringes or drugs used according to study group. Group A: 5 mg Remifentanyl in 50 cc (100 ug/ml). Bolus of 2 ug/kg IBW (0,2 ml / 10 kg IBW) followed by 10 - 50 ug/kg IBW/h (1 - 5 ml / 10 kg IBW / h) Group B: Sevoflurane inhalation 1 MAC in O2/air Group C: 200 mg rocuronium in 20 cc (10 mg/ml). Bolus of 1 ml / 10 kg IBW followed by 1 ml / 10 kg IBW/h

Anesthesia will be maintained with Propofol infusion at 5 - 10 mg/kg IBW/hour, lidocaine at 0,75 - 2,25 mg/kg IBW/h, Dexmedetomidine 0,5 - 1,4 ug/kg IBW/h and Ketamine 0,125 - 0,375 mg/kg IBW/h adapted according to Bispectral analysis (BIS) value ( keep below 60) and hemodynamic parameters (keep heart rate below 100 and SAP below 140mmHg).

Maximum infusion rate for propofol: 10 mg/kg/h; for lidocaine 3 mg/kg/h; for ketamine 0,5 mg/kg/h and for dexmedetomidine 1,4 mg/kg/h.

All patients will be ventilated with O2/air and a positive end expiratory pressure (PEEP) > 7 to an end tidal CO2 below 35 mmHg to prevent diaphragmatic activation.

A verres needle will be placed minimum 15 minutes after induction. If the surgeon is not able to place the verres needle in two attempts, every patient will be given a rocuronium bolus of 0.6 mg/kg IBW and the surgeon is asked after 5 minutes to repeat the trocar positioning. This will be noted as a failure to position the verres needle and to inflate the abdomen.

When the abdomen is inflated the first trocar is placed and the positions of the trocar and gastric tube verified, and the stomach confirmed to be empty.

The first abdominal pressure volume relation (APVR) will be measured using the following procedure by the surgeon:

1. The abdomen is deflated of all air by manual palpation of the abdomen and turning the trocar. The abdomen is re-inflated successively to 0.5, 1, 1.5, and 2 liters (IAV), and, at each volume, the intra-abdominal pressure (IAP) is measured while inflation is stopped. A maximum pressure of 15 mmHg is used. The lowest IAP or end expiration value is taken. This allows the drawing of the first APVR, the calculation of the E, PV0, and inflated volume at 15 mmHg.
2. At the end of insufflation, the insufflator is stopped and the insufflation line is closed with a clamp. The IAP is recorded while pressure stabilizes. If no stabilization is achieved in 15 seconds, a leak is possible and the patient is not included in the study or the step-wise inflation is repeated after the leak is closed.

Breathing against the ventilator or pressing is diagnosed when the IAP rises 5 mmHg above the set pressure not by a surgical act, when capnography shows irregularities in the waveform, or when the respiratory rate is higher than the set value. These patients are not included in the randomisation.

All remaining patients will be randomly assigned to three groups. A randomization number will be generated by the secretary of anesthesia at the moment of the patient's enrollment, using a random number generator. The anesthesiologist will be informed of the number when ready to prepare the drugs available from the pharmacy.

The anesthesiologist will not be blinded (i.e., he/she will know what drug he/she gives), because the administration routes are different: iv infusion, iv bolus, or inhalation. The surgeon and OR nurses will be blinded to the drugs used as iv infusion and bolus will always be given.

Group A: A bolus of remifentanyl 2 µg/kg IBW (0,2 ml/ 10 kg IBW) will be given and followed by 10 - 50 ug/kg IBW/h remifentanyl infusion (1 - 5 ml / 10 kg IBW / h). The propofol and dexmedetomidine infusion will be continued but adapted in dose when needed after the measurements.

Group B: Desflurane inhalation at 1 MAC N2/O2 will be started with a fresh gas flush of the ventilator ( using et tidal control function) until the end tidal concentration reaches 1 MAC while the propofol infusion is stopped. The Ketamine Lidocaine Dexmedetomidine infusion is continued.

Group C: A bolus dose of rocuronium 1 mg/kg IBW will be given while the propofol and Dexmedetomidine infusion is continued.

After the above drugs are administered, there will be a waiting period of 5 minutes while the abdomen remains deflated in all groups. The BIS value should stay below 40% in all groups until the second APVR is measured, using the same setup as the first measurement.

After the second APVR measurement the pressure needed to reach 4 liter is calculated and the insufflator is set to this value with a maximum of 15 mmHg in every patient. If during the second APVR the patient presses or breathes against the ventilator this will be noted as a failure to measure the APVR. A dose of rocuronium 1 mg/kg IBW is given followed by an infusion to keep PTC < 4.

The anesthesia is continued with propofol/remifentanyl/Dex in group A, with sevoflurane/Dex in group B, and with Propofol/Dex/Rocuronium in group C. A bolus of sufentanil can be added in any patient after the two APVR measurements, at the discretion of the anesthesiologist.

The surgeon is asked 5 minutes after second APVR if he has sufficient workspace to reach all places he need to operate. He is asked to grade this on a scale of 1 to 5, with 5 excellent and 1 impossible. If the grade is less than 3 and patient didn't get yet any NMB until that time a bolus of rocuronium 1 mg/kg IBW is given. The NMB will be kept in these patients at train of four (TOF) = 0 and PTC < 4 until release of the pneumoperitoneum.

A reversal with 4 mg/kg sugammadex will be given before awakening the patient. Any inadvertent event will be noted. TOF monitoring will be used in all patients to verify when and how deep NMB is given and to verify that sugammadex returns the TOF to a minimum of 90%.

An external statistical group revealed that an enrollment of 12, 14 and 16 patients in the first, second and third group would be sufficient. The difference between the three groups is due to the fact that a comparison is needed between NMB and the other drugs, not between remifentanyl and sevoflurane.

A two way Anova will be used to evaluate the different effect of remifentanyl, sevoflurane versus rocuronium on the abdominal workspace (pressure needed to achieve 4 l) and on the surgical incidence of having an insufficient workspace. ( 2 independent variables, three conditions)

ELIGIBILITY:
Inclusion Criteria:

1. Laparoscopic bariatric surgery in a patient older than 18 years of age without previous laparotomy. Examples of laparoscopic bariatric procedures are gastric band, sleeve gastrectomy, gastric bypass, gastric bypass after lap band, and revision of a gastric bypass

Exclusion Criteria:

1. Allergies or contraindications to the use of one or more of the following drugs: propofol, rocuronium, sugammadex, remifentanyl, or sevoflurane
2. History of a laparotomy
3. Emergency laparoscopy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan P Mulier, PhD, Principal Investigator — azsintjan
Locations (1):
- Azsintjan, Bruges, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study is performed in operating theatre of one center: and one campus: campus Brugge, center: AZ SINT JAN Brugge-Oostende. study is performed on patients requiring laparoscopy for bariatric surgery.
Pre-assignment Details: 8 patients were excluded from randomization due to movements and impossibility to measure abdominal compliance before randomization.
Period: Overall Study
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl
Started | 16 | 14 | 12
Completed | 16 | 14 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl | Total
Number analyzed (Participants) | 16 | 14 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 12 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — the is the age of the patients recorded in number of years.
  years | 38.93 (5.54) | 36.5 (8.4) | 40.67 (7.33) | 38.61 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 9 | 31
  Male | 4 | 4 | 3 | 11
Region of Enrollment [Number; unit: participants]
  Belgium | 16 | 14 | 12 | 42
Elastance [Mean (Standard Deviation); unit: mmHg/Liter] — Elastance: change in pressure (mmHg) for a change in volume (L)
  mmHg/Liter | 2.66 (1.38) | 2.57 (1.44) | 2.58 (1.0) | 2.61 (1.05)
PV0 [Mean (Standard Deviation); unit: mmHg] — pressure at zero volume Measure Description: abdominal pressure at zero volume (PV0) pressure is measured by pressure transducer in insufflator PVO is measured as the initial pressure before insufflation starts
  mmHg | 7.3 (3.37) | 7.9 (3.37) | 6.5 (1.5) | 7.4 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Anesthetics on the Pressure at Zero Volume (PV0) Measured During Insufflation of the Abdomen
Description: the impact of the following agents on the pressure at zero volume (PV0): remifentanyl > 0.50 µg/kg/min; sevoflurane 1 MAC and deep neuromuscular block (rocuronium given with PTC < 4).
Time Frame: 5 min after reaching 1 MAC or haven given the anesthetics intravenous
Population: laparoscopic bariatric surgery population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl
Number analyzed (Participants) | 16 | 14 | 12
mmHg | 5.7 (1) | 8.29 (3.6) | 6.58 (1.39)

2. Primary Outcome: Effect of Anesthetics on the Abdominal Elastance (E) Measured During Insufflation of the Abdomen by
Description: the impact of the following agents on the abdominal elastance (E) : remifentanyl > 0.50 µg/kg/min; sevoflurane 1 MAC and deep neuromuscular block (rocuronium given with PTC < 4).
Time Frame: 5 min after reaching 1 MAC or haven given the anesthetics intravenous
Population: laparoscopic bariatric surgery population
Measure: Mean (Standard Deviation); unit: mmHg/liter
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl
Number analyzed (Participants) | 16 | 14 | 12
mmHg/liter | 2.53 (1.23) | 2.71 (1.44) | 2.5 (0.8)

3. Secondary Outcome: Adverse Events Difference Between the Three Groups
Description: To compare the major adverse events among the patient groups who receive the different agents listed above in the "primary efficacy objective"
Time Frame: from zero till 24 hours after recovery of surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl
Number analyzed (Participants) | 16 | 14 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: one month post operative
Arm/Group | Deep Neuromuscular Block | Inhalation With 1 MAC Sevoflurane | Remifentanyl
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Neuromuscular Block (N=16) | Inhalation With 1 MAC Sevoflurane (N=14) | Remifentanyl (N=12)
post operative bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — post operative hypertension and bleeding requiring admission on intensive care followed by laparoscopic revision for bleeding. patient recovered without any remaining lesions.

LIMITATIONS AND CAVEATS:
Patients with central obesity were not included in this study patients were it was not possible to measure the abdominal compliance without neuromuscular block were not included in this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No